CLINICAL TRIAL: NCT02601157
Title: Harmonizing Optimal Strategy for Treatment of Coronary Artery Stenosis - Coronary Intervention With Next Generation Drug-Eluting Stent Platforms and Abbreviated Dual Antiplatelet Therapy (HOST-IDEA) Trial
Acronym: HOST-IDEA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: B. Braun Korea Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Director of Cardiac Catheterization Laboratory & Coronary Intervention, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOST-IDEA trial
Record Dates: First submitted 2015-11-07; First posted 2015-11-10 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Stable Angina; Unstable Angina; Non-ST Segment Elevation Myocardial Infarction
Keywords: stent; polymer; antiplatelet therapy; clopidogrel
MeSH Terms: conditions — Angina, Stable; Angina, Unstable | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Aspirin; Clopidogrel; Prasugrel Hydrochloride; Ticagrelor; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orsiro SES or CX-ISAR/3-months DAPT (Experimental): Patients allocated to this group will be implanted with Orisro sirolimus-eluting stents or Corflex ISAR stents for their coronary lesions, and then will be followed with 3-month dual antiplatelet therapy (DAPT) schedule.
  Interventions: Drug: 3-months DAPT
- Orsiro SES or CX-ISAR/1-year DAPT (Active Comparator): Patients allocated to this group will be implanted with Orisro sirolimus-eluting stents or Coroflex ISAR stents for their coronary lesions, and then will be followed with 1-year dual antiplatelet therapy (DAPT) schedule.
  Interventions: Drug: 1-year DAPT

INTERVENTIONS:
Drug: 3-months DAPT — Contrast to the conventional 1-year DAPT, patients in this group will be followed with 3-months DAPT schedule after the stenting
  Other Names: Aspirin + P2Y12 inhibitor (clopidogrel/prasugrel/ticagrelor) for 3-months schedule after the coronary stenting
  Arms: Orsiro SES or CX-ISAR/3-months DAPT
Drug: 1-year DAPT — Patients in this group will be followed with the conventional 1-year DAPT schedule after the stenting
  Other Names: Aspirin + P2Y12 inhibitor (clopidogrel/prasugrel/ticagrelor) for 1-year schedule after the coronary stenting
  Arms: Orsiro SES or CX-ISAR/1-year DAPT

SUMMARY:
We had little experience in coronary intervention with recently introduced newer drug-eluting stent (DES) platforms, despite great anticipation, and optimal duration of dual antiplatelet therapy (DAPT) for these stent systems still needs to be established.

Herein, we plan the HOST-coronary intervention with next-generation drug-eluting stent platforms and abbreviated dual antiplatelet therapy (HOST-IDEA) trial to compare single antiplatelet therapy (SAPT) after 3-month DAPT with 12-month DAPT in all-comers undergoing coronary intervention with third-generation DES with the thinnest struts.

P2Y12 inhibitor treatment is added to aspirin during the 3-months period after the stenting, and this abbreviated duration of DAPT will be compared with conventional 1-year mandatory DAPT regimen in a 1:1 randomized stratification.

Net adverse clinical events (NACEs), a composite of cardiac death, target vessel related myocardial infarction, clinically-drivent target lesion revascularization, definite or probable stent thrombosis and major bleeding is a primary endpoint for evaluating safety and efficacy of the difference of DAPT duration.

1-year target lesion failure (TLF) as a composite of cardiac death, target vessel related myocardial infarction and clinically driven target lesion revascularization will be identified as a secondary ischemic outcome. 1-year major bleeding events classified as BARC type 3 or 5 bleeding events will be identified as a secondary bleeding outcome.

With this trial, you will be able to get clear insight on the behavior of newer DES platforms. Reference data for the shortened mandatory DAPT regimen will also be delineated in the selected patients, and it might be helpful to those who need it.

DETAILED DESCRIPTION:
Every antiplatelet-naïve patient undergoing an elective procedure will be given 300 mg aspirin and loading dose of one of P2Y12 receptor inhibitors (e.g., 600 mg clopidogrel, 60 mg prasugrel or 180 mg ticagrelor) preferably ≥2 hours before the intervention. These loading doses can be waived for chronic antiplatelet users, and prasugrel or ticagrelor can be used instead of clopidogrel. Choice for P2Y12 inhibitors will be left to responsible physicians' discretion, and this decision will be based on the patient/lesional characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with de novo stenotic lesions who are suitable for coronary stenting with drug-eluting stent

Exclusion Criteria:

* 1. High risk profiles for ischemic adverse events such as A. ST-segment elevation myocardial infarction (STEMI) B. Patients with cardiogenic shock or concomitant severe decompensated heart failure C. Myocardial infarction or stent thrombosis in spite of the maintenance of antiplatelet therapy D. Restenosis in stented segments or previous sites of balloon angioplasty 2. Patients who cannot follow allocated DAPT schedule due to the planned surgery or elective procedure within 3 months after the stenting 3. Recent history of major surgery or evident events of gastrointestinal bleeding within 1 month from the procedure 4. Patients on anticoagulation therapy with warfarin or other anticoagulants 5. Life expectancy less than 1 year (such as malignancies or other chronic systemic diseases) 6. Pregnant women 7. Past history of allergy or other contraindications for the following medications/materials: aspirin, clopidogrel, heparin, cobalt chromium, sirolimus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2173 (Actual)
Dates: Start 2016-01-18; Primary Completion 2021-08-14 (Actual); Study Completion 2022-08-14 (Actual)

PRIMARY OUTCOMES:
NACEs (net adverse clinical events) | post-stenting 12 months
  a composite of cardiac death, target vessel-related non-fatal myocardial infarction, clinically-driven target lesion revascularization, definite or probable stent thrombosis, and major bleeding

SECONDARY OUTCOMES:
TLF (target lesion failure) | post-stenting 12 months
  a composite of cardiac death, target vessel-related non-fatal myocardial infarction, and clinically-driven target lesion revascularization
Major bleeding | post-stenting 12 months
  Major bleeding events classified as BARC type 3 or 5 bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, M.D., Ph.D., Study Chair — Seoul National University Hospital
Locations (12):
- South Korea (12):
  - Busan Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - SoonChunHyang University Cheonan Hospital, Cheonan
  - Chonnam National University Hospital, Gwangju
  - Gwangju Christian Hospital, Gwangju
  - Ewha Womans University Medical Center Mokdong Hospital, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon

REFERENCES:
- [Derived] Han JK, Hwang D, Yang S, Park SH, Kang J, Yang HM, Park KW, Kang HJ, Koo BK, Hur SH, Kim W, Kim SY, Park SH, Han SH, Kim SH, Shin S, Park K, Lee SJ, Kim JW, Lee N, Kim HS. Abbreviated dual antiplatelet therapy after percutaneous coronary intervention with ultrathin-strut drug-eluting stents in South Korea: 3-year outcomes of the multicentre, randomised HOST-IDEA trial. EClinicalMedicine. 2025 Dec 18;91:103698. doi: 10.1016/j.eclinm.2025.103698. eCollection 2026 Jan. PMID 41509615
- [Derived] Han JK, Lee K, Park SH, Yang S, Hwang D, Kang J, Yang HM, Park KW, Kang HJ, Koo BK, Hur SH, Kim W, Park SH, Han SH, Kim SH, Kim YH, Lee N, Lee SJ, Shin S, Kim HS. Short-Term DAPT After Complex PCI With Third-Generation DES: A Post Hoc Analysis of the HOST-IDEA Trial. Circ Cardiovasc Interv. 2025 May;18(5):e014623. doi: 10.1161/CIRCINTERVENTIONS.124.014623. Epub 2025 Mar 31. PMID 40160090
- [Derived] Han JK, Yang S, Hwang D, Park SH, Kang J, Yang HM, Park KW, Kang HJ, Koo BK, Cho JM, Cho J, Bang DW, Lee JH, Lee HC, Kim KJ, Chun WJ, Seo WW, Park WJ, Park SM, Kim JW, Kim HS. Biodegradable Polymer Versus Polymer-Free Ultrathin Sirolimus-Eluting Stents: Analysis of the Stent Arm Registry From the HOST-IDEA Randomized Trial. Circ Cardiovasc Interv. 2024 Jul;17(7):e013585. doi: 10.1161/CIRCINTERVENTIONS.123.013585. Epub 2024 May 24. PMID 38786579
- [Derived] Han JK, Hwang D, Yang S, Park SH, Kang J, Yang HM, Park KW, Kang HJ, Koo BK, Hur SH, Kim W, Kim SY, Park SH, Han SH, Kim SH, Shin S, Kim YH, Park K, Lee N, Lee SJ, Kim JW, Kim HS. Comparison of 3- to 6-Month Versus 12-Month Dual Antiplatelet Therapy After Coronary Intervention Using the Contemporary Drug-Eluting Stents With Ultrathin Struts: The HOST-IDEA Randomized Clinical Trial. Circulation. 2023 May 2;147(18):1358-1368. doi: 10.1161/CIRCULATIONAHA.123.064264. Epub 2023 Mar 5. PMID 36871230
- [Derived] Kim CH, Han JK, Yang HM, Park KW, Lee HY, Kang HJ, Koo BK, Lee N, Cha TJ, Yang TH, Jeong MH, Yoon MH, Lee SU, Lee SJ, Kim JW, Cho JM, Han KR, Pyun WB, Kim HS. Study protocol for a randomised controlled trial: harmonising optimal strategy for treatment of coronary artery stenosis - coronary intervention with next-generation drug-eluting stent platforms and abbreviated dual antiplatelet therapy (HOST-IDEA) trial. BMJ Open. 2017 Oct 11;7(10):e016617. doi: 10.1136/bmjopen-2017-016617. PMID 29025834